CLINICAL TRIAL: NCT01001078
Title: Prospective Randomized Trial Comparing the Performance of Two Supraglottic Airway Management Devices: I-Gel and Supreme LMA
Brief Title: Comparison Study of Two Supraglottic Airway Devices Used for Patients Under General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Nikola Joly, MD, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: HMR-Anesth-Joly
Record Dates: First submitted 2009-10-21; First posted 2009-10-23 (Estimated); Results first posted 2015-01-22 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Anesthesia Airway Management
Keywords: supraglottic airway devices; I-Gel; Supreme Laryngeal mask airway; Airway leak pressure; peak airway pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- I-Gel supraglottic airway device (Active Comparator): Group in which the I-Gel will be used in the first and second attempts to secure the airway. If a third attempt is needed, the LMA Supreme will be used. If the third attempt fails, a standard endotracheal tube will be used.
  Interventions: Device: I-Gel supraglottic airway device; Device: Standard endotracheal tube
- LMA Supreme supraglottic airway device (Active Comparator): Group in which the LMA Supreme will be used in the first and second attempts to secure the airway. If a third attempt is needed, the I-Gel will be used. If the third attempt fails, a standard endotracheal tube will be used.
  Interventions: Device: LMA Supreme supraglottic airway device; Device: Standard endotracheal tube
- Standard endotracheal tube (Active Comparator): A Standard endotracheal tube will be inserted in case both other airway devices (LMA Supreme and iGel) devices fail to provide adequate ventilation.
  Interventions: Device: Standard endotracheal tube

INTERVENTIONS:
Device: I-Gel supraglottic airway device — 2 attempts to secure the airway will be tried. If they both fail, there will be a crossover with a Supreme LMA.
  Arms: I-Gel supraglottic airway device
Device: LMA Supreme supraglottic airway device — In the LMA Supreme group, the same interventions will be done as in the I-Gel group. The cuff of the LMA Supreme will be inflated with 25 mL of air and then by intervals of 5 mL until no leak is heard (max 45 mL). Leak pressure will also be measure at 45 mL. Once the leak test is done, the cuff will be deflated to initial volume necessary to avoid audible leaks.
  Arms: LMA Supreme supraglottic airway device
Device: Standard endotracheal tube — In case both supraglottic airway devices fail, a standard endotracheal tube will be inserted

SUMMARY:
This study will compare two supraglottic airway devices currently on the market. Supraglottic airway devices are used during general anesthesia to provide a patent airway. They are inserted blindly into the mouth once the patient has lost consciousness and they cover the laryngeal inlet. The I-Gel and the Supreme laryngeal mask airway (LMA) are the two devices to be compared. The I-Gel has no inflatable cuff, which makes it different from all other supraglottic airway devices currently in use. The Supreme shares some characteristics of the other LMA devices, but it is disposable. Our main goal will be to compare the airway leak pressure and the peak airway pressure of each devices. We will also measure the time needed for insertion, number of attempts needed to secure the airway and side effects related to the airway (cough, dysphagia, trauma, hoarseness of voice, sore throat).

DETAILED DESCRIPTION:
First of all, we will record the following demographic variables: age, sex, height, weight, BMI, surgery planned, American Society of Anesthesiology (ASA) status, dental state (good, bad, edentulous), tobacco use (none, ceased, active) and packs year, Mallampati score, thyromental distance and whether or not there is trauma on the tongue, teeth or lips prior to surgery.

Induction of anesthesia will be standardized with Fentanyl 1-3 mcg/kiloGram(kG) and Propofol 1-3,5 mg/kG. The use of myorelaxant will be mandatory, but either succinylcholine or rocuronium will be used as long as complete disappearance of T1 is observed before attempting supraglottic airway insertion.

Prior to insertion, ease of ventilation (yes/no) will be noted.

The two airway devices will be used according to manufacturers instructions. The sizes of the devices will be chosen according to weight:

I-Gel: 50-90 kG: #4 and 90 Kg and up: #5 LMA Supreme: 50-70 Kg: #4 and 70-100 Kg: #5.

Patients will be randomized in either I-Gel or LMA Supreme group. Two insertions with the same device will be allowed before a crossover to the other device. If the third attempt fails, a standard endotracheal tube will be put in the trachea and blood in the oral cavity will be sought. After each failed attempt (no thoracic expansion, no carbon dioxide (CO2) square wave or leak at standardized volume. Blood on the devices will also be recorded.

Since the LMA Supreme has a cuff, we will inflate it to 25 mL and then by intervals of 5 mL of air (max 45 mL) we will inflate it at a volume where no audible leak is heard at a standardized ventilation scheme of volume controlled 8 mL/kg X 10 breaths per minute.

Once fixed with tape, we will measure peak and mean airway pressure for three breaths after 30 seconds of volume controlled breathing. Then the fresh gas flow will be fixed at 3 L/min of 50-50 air-oxygen blend and the Adjustable Pressure Limiting valve will be closed. We will look either for a plateau pressure at which a leak equal to the fresh gas flow or a pressure of 40 cm of water.

We will sought adverse effect like bronchospasm, cough, regurgitation, desaturation, aspiration and deglutition movement.

Ease of insertion will be score on a scale of 1 to 4. 1 being very easy and 4 being very hard.

Endoscopic evaluation will take place afterwards. First in the ventilation tube. Scoring for laryngeal view:

1. Vocal cords all visible;
2. Partial view of the cords including arytenoids;
3. View of the epiglottis only;
4. Other (LMA or pharynx).

Downfolding of the epiglottis will be sought.

Then we will go through the oesophageal port and see if the oesophageal mucosa il visible.

During surgery, we will check if airway manipulation and/or withdrawal was necessary and why.

If traces of blood on the devices are present at the end of the intervention it will be noted.

Two interviews will take place one at the post anesthesia care unit and another the following day by phone if the patient was having ambulatory surgery. Sore throat, cough, dysphagia and dysphonia will be asked to be graded: absent, mild, moderate or severe.

Pulse and arterial pressure with the operating room's sphygmomanometer and oximeter will be written before induction, after induction before insertion and at 1 and 2 minutes post insertion.

ELIGIBILITY:
Inclusion Criteria:

* Weight more than 50 kg;
* Body Mass Index less than 30;
* ASA I to III.

Exclusion Criteria:

* Symptomatic gastro oesophageal reflux disease (GERD);
* Non fasted patients;
* Nasogastric tube in place;
* Intestinal obstruction;
* Ear, nose and throat surgery in the past or deformation of the airway;
* Known difficult airway (Cormack-Lehane grade 3-4);
* Oral cavity opening less than 3 cm;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Drolet, MD, FRCPC, Principal Investigator — Hôpital Maisonneuve-Rosemont, Université de Montréal
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada

REFERENCES:
- [Background] Theiler LG, Kleine-Brueggeney M, Kaiser D, Urwyler N, Luyet C, Vogt A, Greif R, Unibe MM. Crossover comparison of the laryngeal mask supreme and the i-gel in simulated difficult airway scenario in anesthetized patients. Anesthesiology. 2009 Jul;111(1):55-62. doi: 10.1097/ALN.0b013e3181a4c6b9. PMID 19512881
- [Background] Janakiraman C, Chethan DB, Wilkes AR, Stacey MR, Goodwin N. A randomised crossover trial comparing the i-gel supraglottic airway and classic laryngeal mask airway. Anaesthesia. 2009 Jun;64(6):674-8. doi: 10.1111/j.1365-2044.2009.05898.x. PMID 19453322
- [Background] Weber U, Oguz R, Potura LA, Kimberger O, Kober A, Tschernko E. Comparison of the i-gel and the LMA-Unique laryngeal mask airway in patients with mild to moderate obesity during elective short-term surgery. Anaesthesia. 2011 Jun;66(6):481-7. doi: 10.1111/j.1365-2044.2011.06682.x. PMID 21568982
- [Background] Gatward JJ, Cook TM, Seller C, Handel J, Simpson T, Vanek V, Kelly F. Evaluation of the size 4 i-gel airway in one hundred non-paralysed patients. Anaesthesia. 2008 Oct;63(10):1124-30. doi: 10.1111/j.1365-2044.2008.05561.x. Epub 2008 Jul 9. PMID 18616521
- [Background] Richez B, Saltel L, Banchereau F, Torrielli R, Cros AM. A new single use supraglottic airway device with a noninflatable cuff and an esophageal vent: an observational study of the i-gel. Anesth Analg. 2008 Apr;106(4):1137-9, table of contents. doi: 10.1213/ane.0b013e318164f062. PMID 18349185
- [Background] Uppal V, Fletcher G, Kinsella J. Comparison of the i-gel with the cuffed tracheal tube during pressure-controlled ventilation. Br J Anaesth. 2009 Feb;102(2):264-8. doi: 10.1093/bja/aen366. PMID 19151051
- [Background] Wong DT, Yang JJ, Jagannathan N. Brief review: The LMA Supreme supraglottic airway. Can J Anaesth. 2012 May;59(5):483-93. doi: 10.1007/s12630-012-9673-0. Epub 2012 Feb 9. PMID 22318376
- [Background] Keller C, Brimacombe JR, Keller K, Morris R. Comparison of four methods for assessing airway sealing pressure with the laryngeal mask airway in adult patients. Br J Anaesth. 1999 Feb;82(2):286-7. doi: 10.1093/bja/82.2.286. PMID 10365012
- [Background] Brimacombe J, Berry A. A proposed fiber-optic scoring system to standardize the assessment of laryngeal mask airway position. Anesth Analg. 1993 Feb;76(2):457. No abstract available. PMID 8424538
- [Background] Teoh WH, Lee KM, Suhitharan T, Yahaya Z, Teo MM, Sia AT. Comparison of the LMA Supreme vs the i-gel in paralysed patients undergoing gynaecological laparoscopic surgery with controlled ventilation. Anaesthesia. 2010 Dec;65(12):1173-9. doi: 10.1111/j.1365-2044.2010.06534.x. Epub 2010 Oct 19. PMID 20958278
- [Background] Russo SG, Cremer S, Eich C, Jipp M, Cohnen J, Strack M, Quintel M, Mohr A. Magnetic resonance imaging study of the in vivo position of the extraglottic airway devices i-gel and LMA-Supreme in anaesthetized human volunteers. Br J Anaesth. 2012 Dec;109(6):996-1004. doi: 10.1093/bja/aes314. Epub 2012 Sep 25. PMID 23015619
- [Background] Chew EE, Hashim NH, Wang CY. Randomised comparison of the LMA Supreme with the I-Gel in spontaneously breathing anaesthetised adult patients. Anaesth Intensive Care. 2010 Nov;38(6):1018-22. doi: 10.1177/0310057X1003800609. PMID 21226431
- [Background] Ragazzi R, Finessi L, Farinelli I, Alvisi R, Volta CA. LMA Supreme vs i-gel--a comparison of insertion success in novices. Anaesthesia. 2012 Apr;67(4):384-8. doi: 10.1111/j.1365-2044.2011.07002.x. Epub 2012 Feb 13. PMID 22329593
- [Background] Chen X, Jiao J, Cong X, Liu L, Wu X. A comparison of the performance of the I-gel vs. the LMA-Sduring anesthesia: a meta-analysis of randomized controlled trials. PLoS One. 2013 Aug 12;8(8):e71910. doi: 10.1371/journal.pone.0071910. eCollection 2013. PMID 23951266
- [Background] Halwagi AE, Massicotte N, Lallo A, Gauthier A, Boudreault D, Ruel M, Girard F. Tracheal intubation through the I-gel supraglottic airway versus the LMA Fastrach: a randomized controlled trial. Anesth Analg. 2012 Jan;114(1):152-6. doi: 10.1213/ANE.0b013e318236f438. Epub 2011 Nov 10. PMID 22075016
- [Background] Michalek P, Donaldson W, Graham C, Hinds JD. A comparison of the I-gel supraglottic airway as a conduit for tracheal intubation with the intubating laryngeal mask airway: a manikin study. Resuscitation. 2010 Jan;81(1):74-7. doi: 10.1016/j.resuscitation.2009.10.009. Epub 2009 Nov 17. PMID 19926388
- [Background] Hernandez MR, Klock PA Jr, Ovassapian A. Evolution of the extraglottic airway: a review of its history, applications, and practical tips for success. Anesth Analg. 2012 Feb;114(2):349-68. doi: 10.1213/ANE.0b013e31823b6748. Epub 2011 Dec 16. PMID 22178627
- [Derived] Joly N, Poulin LP, Tanoubi I, Drolet P, Donati F, St-Pierre P. Randomized prospective trial comparing two supraglottic airway devices: i-gel and LMA-Supreme in paralyzed patients. Can J Anaesth. 2014 Sep;61(9):794-800. doi: 10.1007/s12630-014-0198-6. Epub 2014 Aug 21. PMID 25141831

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was done at a university hospital mainly in the ambulatory surgery unit from september 2009 to april 2011. 50 patients were recruited in 2009, one fourth in 2010 and the last fourth in 2011. 311 patients were assessed for eligibility, 211 were excluded. 178 did not meet inclusion criteria and 33 declined to participate.
Groups:
- I-Gel: Group in which the I-Gel will be used in the first and second attempts to secure the airway. If a third attempt is needed, the LMA Supreme will be used. If the third attempt fails, a standard endotracheal tube will be used.
  Peak and mean airway pressure will be measured once the device is fixed with tape to the patient. Leak pressure will be measured as well. It will be done while closing the Adjustable Pressure Limiting valve and putting the fresh gas flow at 3 L/min. We will be looking at the manometer to see either a plateau (that would be a leak equal to the fresh gas flow) or the maximum allowed pressure 40 cm H2O.
- LMA Supreme: Group in which the LMA Supreme will be used in the first and second attempts to secure the airway. If a third attempt is needed, the I-Gel will be used. If the third attempt fails, a standard endotracheal tube will be used.
  The cuff of the LMA Supreme will be inflated with 25 mL of air and then by intervals of 5 mL until no leak is heard (max 45 mL). Peak and mean airway pressure will be measured once the device is fixed with tape to the patient. Leak pressure will be measured at a cuff volume without audible leak and also at 45 mL. It will be done while closing the Adjustable Pressure Limiting valve and putting the fresh gas flow at 3 L/min. We will be looking at the manometer to see either a plateau (that would be a leak equal to the fresh gas flow) or the maximum allowed pressure 40 cm H2O. Once the leak tests are done, the cuff will be deflated to initial volume necessary to avoid audible leaks.
Period: Overall Study
Arm/Group | I-Gel | LMA Supreme
Started | 50 | 50
Received Allocated Intervention | 46 | 46
Received Crossover | 2 | 3
Intubated | 2 | 1
Lost to Followup Interview | 5 (Could not be interviewed.) | 2 (Could not be interviewed.)
Completed | 50 (Analyzed: 46, excluded from interview analysis: 5) | 50 (Analyzed: 46, excluded from interview analysis: 2)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Since previous studies on SAD had found SD values for leak pressure around seven cmH2O, it was estimated that fifty patients per group would allow us to find a difference just under four cmH2O between groups with an alpha error = 0.05 and a power of 80%.
Groups:
- Total: Total of all reporting groups
Arm/Group | I-Gel | LMA Supreme | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (16) | 50 (18) | 50 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 37 | 70
  Male | 17 | 13 | 30
Weight [Mean (Standard Deviation); unit: kilograms] | 72 (11) | 71 (13) | 71.5 (12)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26 (4) | 26 (4) | 26 (4)
Height [Mean (Standard Deviation); unit: meters] | 1.68 (0.09) | 1.67 (0.10) | 1.68 (0.095)

OUTCOME MEASURES:

1. Primary Outcome: Measure of the Airway Leak Pressure
Time Frame: After introduction of the supraglottic device before the beginning of the surgery.
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | I-Gel | LMA Supreme
Number analyzed (Participants) | 46 | 46
cmH2O | 23 (7) | 21 (8)

2. Secondary Outcome: Measure of the Peak Airway Pressure
Time Frame: After introduction of the SAD before the beginning of the surgery.
Measure: Mean (Standard Deviation); unit: cm H20
Groups:
- I-Gel: Group in which the I-Gel will be used in the first and second attempts to secure the airway. If a third attempt is needed, the LMA Supreme will be used. If the third attempt fails, a standard endotracheal tube will be used.
- LMA Supreme: Group in which the LMA Supreme will be used in the first and second attempts to secure the airway. If a third attempt is needed, the I-Gel will be used. If the third attempt fails, a standard endotracheal tube will be used.
Arm/Group | I-Gel | LMA Supreme
Number analyzed (Participants) | 46 | 46
cm H20 | 14 (3) | 14 (5)

3. Secondary Outcome: Time Needed to Secure the Airway
Time Frame: From opening of the mouth to thoracic expansion and presence of End Tidal CO2 up to five minutes.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | I-Gel | LMA Supreme
Number analyzed (Participants) | 46 | 46
seconds | 19 (7) | 27 (17)

4. Secondary Outcome: Number of Participants With Successful Attempts to Introduce the Devices
Time Frame: At the beginning of anesthesia before the beginning of the surgery.
Measure: Number; unit: participants
Arm/Group | I-Gel | LMA Supreme
Number analyzed (Participants) | 50 | 50
participants
  1st attempt successful | 43 | 44
  2nd attempt successful | 3 | 2
  Crossover device | 2 | 3
  Intubation | 2 | 1

5. Secondary Outcome: Adverse Effects After Anesthesia (Sore Throat, Cough, Dysphagia, Dysphonia)
Description: Intent to treat assessment of adverse events, per intervention, was intended. The adverse effects were assessed by phone; or in person if patient in the hospital; on the following day.
Time Frame: On the day following surgery
Population: 5 participants were lost to follow-up and 4 participants had the crossover device or were intubated in the I-Gel group.
  4 participants were lost to follow-up and 3 participants had the crossover device or were intubated in the LMA Supreme group (one of participants was lost to follow-up and had the crossover device or was intubated)
Measure: Number; unit: participants
Arm/Group | I-Gel | LMA Supreme
Number analyzed (Participants) | 41 | 44
participants
  Sore Throat (absent) | 23 | 26
  Sore Throat (mild) | 10 | 13
  Sore Throat (moderate) | 6 | 4
  Sore Throat (severe) | 2 | 1
  Cough (absent) | 36 | 38
  Cough (mild) | 5 | 5
  Cough (moderate) | 0 | 1
  Cough (severe) | 0 | 0
  Dysphagia (absent) | 25 | 29
  Dysphagia (mild) | 7 | 9
  Dysphagia (moderate) | 9 | 4
  Dysphagia (severe) | 0 | 2
  Dysphonia (absent) | 34 | 35
  Dysphonia (mild) | 5 | 5
  Dysphonia (moderate) | 1 | 3
  Dysphonia (severe) | 1 | 1

6. Secondary Outcome: Airway Manipulation and Blood on Device at Removal
Time Frame: During and after anesthesia when the device is removed.
Measure: Number; unit: participants
Arm/Group | I-Gel | LMA Supreme
Number analyzed (Participants) | 46 | 46
participants
  Repositionning during surgery | 2 | 3
  Blood on device at removal | 5 | 6

ADVERSE EVENTS:
Time Frame: 24 hour after placement of the device
Arm/Group | I-Gel | LMA Supreme
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 23/50 | 31/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | I-Gel (N=50) | LMA Supreme (N=50)
severe sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) — Sore throat graded 4 on a 4-point Likert scale as follows: absent, mild, moderate or severe.
severe cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) — Cough graded 4 on a 4-point Likert scale as follows: absent, mild, moderate or severe.
severe dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) — dysphagia graded 4 on a 4-point Likert scale as follows: absent, mild, moderate or severe.
severe dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — dysphonia graded 4 on a 4-point Likert scale as follows: absent, mild, moderate or severe.
mild sore throat (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 13 (13) — Sore throat graded 2 on a 4-point Likert scale as follows: absent, mild, moderate or severe.
moderate sore throat (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4) — Sore throat graded 3 on a 4-point Likert scale as follows: absent, mild, moderate or severe.
mild dysphagia (Gastrointestinal disorders) | 7 (7) | 9 (9) — Dysphagia graded 2 on a 4-point Likert scale as follows: absent, mild, moderate or severe.
moderate dysphagia (Gastrointestinal disorders) | 9 (9) | 4 (4) — dysphagia graded 3 on a 4-point Likert scale as follows: absent, mild, moderate or severe.
mild dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5) — mild dysphonia graded 2 on a 4-point Likert scale as follows: absent, mild, moderate or severe.
moderate dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) — moderate dysphonia graded 3 on a 4-point Likert scale as follows: absent, mild, moderate or severe.
mild cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5) — mild cough graded 3 on a 4-point Likert scale as follows: absent, mild, moderate or severe.
moderate cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — moderate cough graded 3 on a 4-point Likert scale as follows: absent, mild, moderate or severe.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes